CLINICAL TRIAL: NCT02510677
Title: Three-dimensional Assessment of Intraventricular Dyssynchrony Using Fast Dobutamine Gated SPECT
Acronym: FAST DOGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-176
Record Dates: First submitted 2015-07-22; First posted 2015-07-29 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- myocardial perfusion scintigraphy (Other): Low-dose dobutamine gated SPECT and CZT camera for the assessment of parameters of left ventricular dyssynchrony in heart failure patients eligible for the implantation of a cardiac resynchronization device.
  Interventions: Other: myocardial perfusion scintigraphy

INTERVENTIONS:
Other: myocardial perfusion scintigraphy

SUMMARY:
The prognosis of patients with heart failure has improved due to recent breakthrough in medical treatment and cardiac resynchronization devices. However, there is no paraclinical parameter to assess response to cardiac resynchronization therapy (CRT). This is a major issue since about a third of implanted patients will not be improved by CRT. CZT SPECT allows to perform myocardial perfusion imaging in less than 4 minutes and is able to study myocardial perfusion, viability, left ventricular function, but also ventricular asynchrony.

Using low-dose dobutamine gated SPECT and CZT camera, we aimed to assess left ventricular dyssynchrony in viable segments in patients with heart failure eligible for CRT.

ELIGIBILITY:
Inclusion Criteria:

* Patient with heart failure on optimal medical therapy and targeted for cardiac resynchronization therapy according to current recommendations;
* Age over 18 years
* Clinically stable (without hospitalization for heart failure in the last month)
* Sinus rhythm
* Social security insurance
* Signed consent form

Exclusion Criteria:

* Recent history (less than 21 days) of acute coronary syndrome or unstable angina;
* Recent history (less than 1 month) of acute heart failure;
* Right bundle branch block;
* Irregular heart rate;
* Double-chamber cardiac pacemaker
* Patients previously implanted with a single-chamber cardioverter-defibrillator must have at least 99 percent of unstimulated QRS.
* Countraindication to dobutamine therapy;
* Valvular heart disease, congenital heart disease, hypertrophic cardiomyopathy;
* Significant Ventricular arrhythmias;
* Hypertension (upper than 160/100 mmHg);
* Pregnant, breastfeeding or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
measures of dyssynchrony parameters | baseline
  The primary endpoint is reproducible quantitative measures of dyssynchrony parameters between two successive acquisitions basal (entropy, bandwidth, standard deviation phase histogram).

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine Nucléaire du CHU de Caen, Caen, France